CLINICAL TRIAL: NCT02869048
Title: Amyotrophic Lateral Sclerosis and the Innate Immune System
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Zealand University Hospital (Other); Bispebjerg Hospital (Other); Aarhus University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Anne-Lene Kjældgaard, Ph.d.-student, MD, Rigshospitalet, Denmark
Other Study IDs: H-16017145
Record Dates: First submitted 2016-06-28; First posted 2016-08-16 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Amyotrophic Lateral Sclerosis; Neurodegenerative Disease; Motor Neuron Disease
Keywords: Biological Specimen Banks; Innate Immunity; Clinical Study; Complement system proteins; Amyotrophic lateral sclerosis; Neurodegenerative disease; Motor neuron disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, EDTA-plasma, Hirudin-plasma, Heparin-plasma and RNAlater samples (with fullblood) will be kept in biobank as well as analyzed according design and methods of Clinical study 1+2+3.
  Spinal liquid sample will also be kept in biobank (Clinical Study 2+3).
  10 muscle biopsies from ALS patients will be analyzed (Clinical study 4)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- ALS patients: Patients diagnosed with ALS will be included in this group. Blood and spinal fluid samples will be stored in biobank and later analyzed. A subset of this group (20 ALS patients) will give blood and spinal fluid every 6 months during progression of the disease. A subset of 10 will donate a muscle biopsy.
- Control group with patients with other neurological disease: Patients referred to hospital with symptoms of acute or chronic headache.
- Neurologically healthy control group: Patients having orthopaedic surgery performed in spinal anaesthesia.

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is an aggressive, deadly disease. ALS leads to destruction of the neural pathways which control the conscious movements of the muscles. This destruction leads to muscular dystrophy with increasing difficulties in moving, breathing, swallowing, and speaking. In the last phase of an ALS patient's life it is necessary with respiratory therapy in order to breathe. In average an ALS patient lives 3 years from the time he or she gets the diagnose.

The cause of the disease is still unknown and there is currently no treatment which can stop the progression of the disease. Former clinical studies have indicated that the innate immune system and in particular the complement system plays a significant role in the progression of ALS. The complement system, which is activated in cascades, is part of the innate system but participates in the innate as well as the acquired immune system. Former clinical trials have been characterized by limited knowledge about both the complement system as well as to how it is measured.

Today it is possible to measure directly on the different components of the complement system and to understand its contribution to the overall immune response. It is also possible today to detect defects of the complement system. All these progressions are the foundation for this project which is carried out in close cooperation with one of the world's leading researchers in the complement system, professor Peter Garred from Rigshospitalet.

The aim is to make a national research project about ALS in order to investigate the role of the innate immune system, and especially the complement system, in patients with ALS.

In the long term the hope is, that this will lead the way to a targeted and effective medical treatment to the people affected by this grave disease.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a progressive, deadly, neurodegenerative disease which affects the upper and lower motor neurons. This leads to profound muscular dystrophy, hyperreflexia, fasciculations and paresis of the bulbar as well as the skeletal musculature. ALS causes increasing physical fatigue and the patients soon become bedridden and respiratory insufficient.The diagnosis ALS is made according to the El Escorial revisited. Often clinical and neurophysiological tests must be repeated (1-4).

In Denmark the incidence of ALS is 1-2/100.000 and the prevalence is 4-6/100.000. The average survival time from the time of the diagnosis is 3 years but with great variance. (5+6)

Today the pathogenesis is still unknown and no treatment can stop the progression of ALS. Treatment with riluzole seems to prolong the median time of survival for 2 or 3 months (7).

Most likely, a future medical treatment requires a better understanding of the pathogenesis as well as the pathophysiology of ALS. This present study aims to do so based on the hypothesis that ALS partially or fully is caused by complement activation.

The complement system is a complex system consisting of proteins in plasma as well as membrane bound proteins which together complement the antibody-based immune system. The complement system is a self-perpetuating cascade system which is activated through different pathways. It works by opsonisation where complement proteins bind to microorganisms to activate and target granulocytes, monocytes and macrophages. The complement system also causes cytolysis of microorganisms via MAC (membrane attack complex) by activation of the mast cells. It also inactivates and eliminates burned out immune complexes as well as performing apoptotic renovation.

A recent pilot study of Neuromyelitis Optica has shown how the complement system play a central part in the pathogenesis of a disease that previously was wrongfully perceived as an early stage of Disseminated Sclerosis. These findings resulted in medical treatment with anticomplement (equlizumab) with promising results (8). It is possible that similar pathogenetic mechanisms could be the molecular basis of ALS.

Different research groups have tried to illuminate how the immune system is involved in the progression of ALS (9-35). Several studies support the hypothesis that the complement system is of crucial importance for the onset and progression of ALS. (9-28)

In several clinical trials with ALS plasma it is concluded that ALS plasma is cytotoxic when incubated with healthy red blood cells or healthy nerve tissue. Some research indicates that the cytotoxicity is caused by the complement system. The results cannot, however, be reproduced consequently in all clinical trials. These trials were conducted decades ago where the methods of detecting complement activity were limited. (9-14)

Several animal trials indicate that ALS starts in the neuromuscular junctions (NMJ) and therefore should be considered a distal axonopathy rather than a central neurological disease, which today is the general perception of ALS. (27-31)

The purpose of the project The aim is to increase the knowledge of the pathophysiology of the disease ALS as this possibly may lead us closer to a targeted medical treatment.

The project group wants to investigate if a previously found, unique cytotoxicity in the ALS plasma can be retrieved (9-14). If this is the case, then the modern methods of today make it possible to detect whether the immune system in general, and in particular the complement system, is causing this cytotoxicity.

The establishment of a national research project about ALS and the complement system by making a research biobank with systematically collected blood and spinal liquid from ALS patients from all over the country will ensure the opportunity to find out if the complement system plays a role in the onset and progression of ALS.

Furthermore a pilot study will be conducted with the purpose to investigate if there is complement activity in the NMJ in patients with ALS as it has been shown in a study of ALS mice. (28)

The hypotheses

1. ALS is characterized by an abnormal immune response with cytotoxicity and increased complement activity in plasma which is revealed by the following:

   1. Plasma from patients with ALS shows increased haemolytic activity when incubated with red blood cells from healthy subjects.
   2. The complement activity is increased in the plasma from ALS patients compared with plasma from neurologically healthy subjects and subjects with other neurological disease.
   3. The haemolytic activity in the plasma from ALS patients is correlated with the complement activity.
2. Spinal liquid from ALS patients contains increased complement activity compared with spinal liquid from neurologically healthy subjects and from subjects with other neurological disease.

Patients, materials and methods:

Clinical trial 1(CT1): Haemolytic activity and the complement system in ALS plasma

Number of subjects: 25 patients with ALS, 25 patients with other neurological disease, 25 healthy volunteers

The course of CT1: A blood sample is taken from each patient. The red blood cells and the liquid part of the blood, the plasma, are separated. The red blood cells from different subjects are incubated in an other subjects plasma.The same trial course is repeated after inactivation of the present complement system both by heat and by anti-complement.

Clinical trial 2(CT2): Case-control study aiming to mapping the complement system

Number of subjects:100 patients with ALS, 100 patients with other neurological disease and 100 neurologically healthy patients

The course of CT2:Blood samples and cerebrospinal fluid are prepared and then freezed in a research biobank. Then the samples from the 3 groups of subjects are analysed and compared focusing on the complement system: The complement activation potential is measured in the biological material. A cytokine profile is made as well as mapping the acute phase reactants by multiplex assays. Furthermore the RNA expression profile is made on a cell pellet stabilised with RNA later.

Clinical trial 3(CT3): The complement system of ALS patients over time - a cohort study Number of subjects:20 patients with ALS (subset from CT2)

The course of CT3: Every sixth month the course from the CT2 is repeated. The activity of the complement system in each patient with ALS is analyzed as the disease progresses.

Clinical trial 4(CT4): Searching for complement activity in the NMJ of ALS patients

Number of subjects:10 patients with ALS

The course of CT4: The muscle biopsies are taken and immediately brought to the Dep. of Pathology at Rigshospitalet. Then thin layers of tissue are stained in order to analyze the muscle fibers and the NMJ as well as detecting presence of complement activity.

Conducting the study The project consists of four clinical trials. Inclusion of the subjects is done together with staff in ALS outpatient clinics at hospitals all over the country and subjects for the control groups are included according to the list of inclusion sites below.

Inclusion sites:

ALS outpatient clinic, Neurological clinic, Rigshospitalet Glostrup (CT1+2+3+4) Contact: Chief physician Elisabeth Elmo Neurological Clinic, Rigshospitalet Glostrup (neurological control group, CT1+2) Contact: Professor, Chief physician, dr.med. Rigmor Højland Jensen Neurosurgical Clinic, Rigshospitalet (neurological control group, CT2) Contact: Professor, chief physician, dr.med. Marianne Juhler ALS outpatient clinic, Neurological Dep., Bispebjerg Hospital (CT2) Contact: Chief physician Merete Karlsborg ALS outpatient clinic, Neurological Dep., Roskilde Hospital (CT2 + 3) Contact: Chief physician Helle Thagesen ALS outpatient clinic, Neurological Dep., Odense University Hospital (CT2) Contact: Chief physician, dr.med. Matthias Bode ALS outpatient clinic, Neurological Dep., Aarhus Hospital, Nørrebrogade (Clinical Trial 2) Contact: Chief Physician, ph.d. Anette Torvin Gildhøj Private Hospital, Brøndby (Neurologically healthy control group, Clinical Trial 2) Contact: Anaesthesiologist Niels Anker Pedersen

Power calculations CT1: Haemolytic activity and the complement system in ALS plasma The study Overgaard et al. (18) found a mean difference of about 0,20 (SE 0,052 in the ALS group, N=20, SD 0,22) in the absorbance (415 nm and 5 hours of incubation) between ALS patients and healthy bioanalysts. With α=0,05 og beta=0,20 corresponding to power 0,80 we need to include 21 subjects. As possible drop outs and technically failed are considered tests the investigators choose to include 25 subjects in each group. (36)

CT2: Case-control study mapping the complement system The number of subjects in each group is in this case-control study calculated with α=0,05 The investigators compare the complement activation potential of 3 groups with same amount of subjects in each. In healthy subjects the complement activation potential is 100 % with a normal area ranging from 50-150 % and where the prevalence of low complement activation potential (under 50 %) is under 10 %. With power =0,80 it is calculated to be necessary to include 100 subjects in each group. Hereby it is possible to find statistically significant differences between the groups corresponding to an odds ratio of 2,3, which would correspond to 20 % of ALS patients having a low complement activation potential caused by increased complement activity. (36)

CT3: The complement system of ALS patients over time - a cohort study This is a hypothesis generating study. It is expected that the included 20 ALS patients in this cohort will be a subset from Clinical Trial 2. As a control group at baseline the neurologically healthy control group from Clinical Trial 2 will be used.

CT4: Searching for complement activity in the NMJ of ALS patients There is no previous studies describing the complement activity in the NMJ in living humans. It is therefore not relevant to make a calculation of power.

Data processing CT1: Haemolytic activity and the complement system in ALS plasma Comparing the degree of haemolysis between the ALS patients and the control groups t-test and one way ANOVA are used. For calculating the cut-off values the investigators use receiver operating characteristic (ROC) curves.

CT2: Case-control study mapping the complement system Comparing the concentration of complement and the complement activation potential between ALS patients and the control groups t-test and one way ANOVA are used. In order to calculate the odds for low complement activation potential in the ALS group compared with the control groups the investigators use logistic regression. For calculating the cut-off values receiver operating characteristic (ROC) curves are used.

CT3: The complement system of ALS patients over time - a cohort study As in Clinical Trial 2. Furthermore, regression analysis of the complement activity as a function of time since the onset of ALS, gender, age, subtype of illness and disease progression are conducted.

CT4: Searching for complement activity in the NMJ of ALS patients As in CT2. The degree of complement deposition and muscle pathology is described qualitatively and a blinded scoring in "normal", "light degree" and "severe degree" of changes is conducted. This will be compared quantitatively with 2 x K tables and non-parametric statistics.

Dissemination of results The results of the project will be published in international peer reviewed, journals. Both positive and negative findings will be published.

Perspectivation With the establishment of a big national ALS research biobank it will be possible to conduct many future research projects. Continuous research in ALS is paramount for ALS patients nationally as well as internationally in order to maintain hope for an efficient medical treatment for this aggressive disease is found in the future.

ELIGIBILITY:
Inclusion Criteria:

* For ALS group:Diagnosed with the diagnose category "certain ALS" or "likely ALS according to the El Escorial rev. diagnose criteria
* For Neurological control group: Referred to neurological department to be examined for acute or chronic headache or referred to get a lumbar perfusion test performed.

Exclusion Criteria:

* For all groups (Clinical study 2-3): permanent contraindication for having a lumbar puncture performed
* For Neurological control group: Known with chronic inflammatory disease or autoimmune disease.
* For healthy control group (clinical study 1): Known with any disease
* For healthy control group (clinical study 1): Taking daily medication
* For Neurologically healthy control group (Clinical study 2): Known with neurological disease
* For Neurologically healthy control group (Clinical study 2): Known with chronic inflammatory disease or autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALS group: Patients diagnosed with certain or likely ALS
  Neurological control group:
  Patients being examined for cronical headache or being referred to hospital to get a lumbar perfusion test performed.
  Neurologically healthy control group:
  Clinical study 1: Healty employees from Rigshospitalet Clinical study 2: Neurologically healthy patients having planned orthopaedic surgery performed in spinal anaestesia.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2016-06; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Complement activity | 0-10 year
  The complement activity (measured by haemolytic capacity, complement-activation potential and specific mediators) in ALS patients and compared with 2 control groups.

SECONDARY OUTCOMES:
Subcomponents of the complement cascade | 0-10 years
  If increased complement activity is found, the amount of the different subcomponents of the complement cascade are measured and compared with the 2 control groups.
Inactivation of the complement system | 0-2 years
  The effect of inactivation by heat or inhibition of the complement system with anti-complement in the plasma is analyzed by comparing the degree of haemolysis after incubation compared with the test results of the plasma which is not inactivated by heat nor with added anti-complement.
Indirect profiling of inflammatory proteins present in the blood | 0-10 years
  RNA expression profile of the ALS patients compared with the 2 control groups
Cytokines present in the blood | 0-10 years
  The cytokines are measured in ALS patients and compared with the 2 control groups.
Acut phase reactants | 0-10 years
  The acute phase reactants are measured in ALS patients and compared with the 2 control groups.
Complement activity in the neuromuscular junctions of ALS patients. (Clinical trial 4) | 0-3 years
  The amount of complement deposition as well as complement activity in the neuromuscular junctions are described quantitatively as well as qualitatively
Quantitatively and qualitatively description of ALS muscle fibers. | 0-3 years
  The muscle fibres are described quantitatively as well as qualitatively and compared historically collected material of healthy muscle fibers.
Regression analysis | 0-10 years
  The immune response of the ALS patients is analyzed as a function of sex, age, subtype of disease, stage of disease, severity of disease, duration of disease, present smoking, alcohol consumption, present use of medicine (including riluzole). The regression analysis will be compared when possible with the 2 control groups (sex, age, smoking, alcohol consumption, use of medicine).

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Møller, Prof., MD, Study Chair — Clinic of Neuroanestesiology, Rigshospitalet, Denmark; Peter Garred, Prof., MD, Study Chair — Department of Clinical Immunology; Stephen Wørlich Pedersen, dr.med, Study Chair — Dept. of Neurology, Rigshospitalet Glostrup; Karsten Skovgaard Olsen, Dr.med., Study Chair — Clinic of Neuroanaestesiology, Rigshospitalet Glostrup; Anne Øberg Lauritsen, MD, Study Chair — Clinic of Neuroanaestesiology, Rigshospitalet Glostrup; Eva Løbner Lund, MD, PhD, Study Chair — Dept. of Pathology, Rigshospitalet; Anne-Lene Kjældgaard, MD, Principal Investigator — Clinic of Neuroanaestesiology, Rigshospitalet Glostrup
Locations (8):
- Denmark (8):
  - Dept. of Neurology Aarhus Hospital, Nørrebrogade, Aarhus
  - Gildhøj Private Hospital, Brøndby
  - Clinic of neuroanestesiology, Rigshospitalet Glostrup, Copenhagen
  - Dept. of Neurology, Bisbebjerg Hospital, Copenhagen NV
  - Clinic of Neurosurgery, Rigshospitalet, Copenhagen Ø
  - The Dept. og Neurology, Rigshospitalet Glostrup, Glostrup Municipality
  - Dept. of Neurology, Odense Hospital, Odense C
  - The dept. of Neurology, Roskilde Hospital, Roskilde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen PM, Al-Chalabi A. Clinical genetics of amyotrophic lateral sclerosis: what do we really know? Nat Rev Neurol. 2011 Oct 11;7(11):603-15. doi: 10.1038/nrneurol.2011.150. PMID 21989245
- [Background] Tumer Z, Bertelsen B, Gredal O, Magyari M, Nielsen KC, Lucamp, Gronskov K, Brondum-Nielsen K. Novel heterozygous nonsense mutation of the OPTN gene segregating in a Danish family with ALS. Neurobiol Aging. 2012 Jan;33(1):208.e1-5. doi: 10.1016/j.neurobiolaging.2011.07.001. Epub 2011 Aug 26. PMID 21852022
- [Background] Phukan J, Pender NP, Hardiman O. Cognitive impairment in amyotrophic lateral sclerosis. Lancet Neurol. 2007 Nov;6(11):994-1003. doi: 10.1016/S1474-4422(07)70265-X. PMID 17945153
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847
- [Background] Seals RM, Hansen J, Gredal O, Weisskopf MG. Age-period-cohort analysis of trends in amyotrophic lateral sclerosis in Denmark, 1970-2009. Am J Epidemiol. 2013 Oct 15;178(8):1265-71. doi: 10.1093/aje/kwt116. Epub 2013 Sep 24. PMID 24064744
- [Background] Chio A, Logroscino G, Traynor BJ, Collins J, Simeone JC, Goldstein LA, White LA. Global epidemiology of amyotrophic lateral sclerosis: a systematic review of the published literature. Neuroepidemiology. 2013;41(2):118-30. doi: 10.1159/000351153. Epub 2013 Jul 11. PMID 23860588
- [Background] Annunziata P, Volpi N. High levels of C3c in the cerebrospinal fluid from amyotrophic lateral sclerosis patients. Acta Neurol Scand. 1985 Jul;72(1):61-4. doi: 10.1111/j.1600-0404.1985.tb01548.x. PMID 4050318
- [Background] Apostolski S, Nikolic J, Bugarski-Prokopljevic C, Miletic V, Pavlovic S, Filipovic S. Serum and CSF immunological findings in ALS. Acta Neurol Scand. 1991 Feb;83(2):96-8. doi: 10.1111/j.1600-0404.1991.tb04656.x. PMID 2017904
- [Background] Conradi S, Ronnevi LO. Cytotoxic activity in the plasma of amyotrophic lateral sclerosis (ALS) patients against normal erythrocytes. Quantitative determinations. J Neurol Sci. 1985 May;68(2-3):135-45. doi: 10.1016/0022-510x(85)90095-4. PMID 4009202
- [Background] Conradi S, Ronnevi LO. Immunoglobulin-mediated cytotoxic effect of ALS-plasma towards erythrocytes: reflexion of a pathogenetic mechanism? Adv Exp Med Biol. 1987;209:7-13. doi: 10.1007/978-1-4684-5302-7_2. No abstract available. PMID 3577932
- [Background] Digby J, Harrison R, Jehanli A, Lunt GG, Clifford-Rose F. Cultured rat spinal cord neurons: interaction with motor neuron disease immunoglobulins. Muscle Nerve. 1985 Sep;8(7):595-605. doi: 10.1002/mus.880080709. PMID 4047091
- [Background] Fischer LR, Culver DG, Tennant P, Davis AA, Wang M, Castellano-Sanchez A, Khan J, Polak MA, Glass JD. Amyotrophic lateral sclerosis is a distal axonopathy: evidence in mice and man. Exp Neurol. 2004 Feb;185(2):232-40. doi: 10.1016/j.expneurol.2003.10.004. PMID 14736504
- [Background] Frey D, Schneider C, Xu L, Borg J, Spooren W, Caroni P. Early and selective loss of neuromuscular synapse subtypes with low sprouting competence in motoneuron diseases. J Neurosci. 2000 Apr 1;20(7):2534-42. doi: 10.1523/JNEUROSCI.20-07-02534.2000. PMID 10729333
- [Background] Goldknopf IL, Sheta EA, Bryson J, Folsom B, Wilson C, Duty J, Yen AA, Appel SH. Complement C3c and related protein biomarkers in amyotrophic lateral sclerosis and Parkinson's disease. Biochem Biophys Res Commun. 2006 Apr 21;342(4):1034-9. doi: 10.1016/j.bbrc.2006.02.051. Epub 2006 Feb 20. PMID 16516157
- [Background] Grewal RP, Morgan TE, Finch CE. C1qB and clusterin mRNA increase in association with neurodegeneration in sporadic amyotrophic lateral sclerosis. Neurosci Lett. 1999 Aug 13;271(1):65-7. doi: 10.1016/s0304-3940(99)00496-6. PMID 10471215
- [Background] Heurich B, El Idrissi NB, Donev RM, Petri S, Claus P, Neal J, Morgan BP, Ramaglia V. Complement upregulation and activation on motor neurons and neuromuscular junction in the SOD1 G93A mouse model of familial amyotrophic lateral sclerosis. J Neuroimmunol. 2011 Jun;235(1-2):104-9. doi: 10.1016/j.jneuroim.2011.03.011. Epub 2011 Apr 17. PMID 21501881
- [Background] Kawamata T, Akiyama H, Yamada T, McGeer PL. Immunologic reactions in amyotrophic lateral sclerosis brain and spinal cord tissue. Am J Pathol. 1992 Mar;140(3):691-707. PMID 1347673
- [Background] Kong J, Xu Z. Massive mitochondrial degeneration in motor neurons triggers the onset of amyotrophic lateral sclerosis in mice expressing a mutant SOD1. J Neurosci. 1998 May 1;18(9):3241-50. doi: 10.1523/JNEUROSCI.18-09-03241.1998. PMID 9547233
- [Background] Lee JD, Kamaruzaman NA, Fung JN, Taylor SM, Turner BJ, Atkin JD, Woodruff TM, Noakes PG. Dysregulation of the complement cascade in the hSOD1G93A transgenic mouse model of amyotrophic lateral sclerosis. J Neuroinflammation. 2013 Sep 26;10:119. doi: 10.1186/1742-2094-10-119. PMID 24067070
- [Background] Liveson J, Frey H, Bornstein MB. The effect of serum from ALS patients on organotypic nerve and muscle tissue cultures. Acta Neuropathol. 1975 Aug 11;32(2):127-31. doi: 10.1007/BF00689566. PMID 1166766
- [Background] Lobsiger CS, Boillee S, Cleveland DW. Toxicity from different SOD1 mutants dysregulates the complement system and the neuronal regenerative response in ALS motor neurons. Proc Natl Acad Sci U S A. 2007 May 1;104(18):7319-26. doi: 10.1073/pnas.0702230104. Epub 2007 Apr 26. PMID 17463094
- [Background] Lobsiger CS, Boillee S, Pozniak C, Khan AM, McAlonis-Downes M, Lewcock JW, Cleveland DW. C1q induction and global complement pathway activation do not contribute to ALS toxicity in mutant SOD1 mice. Proc Natl Acad Sci U S A. 2013 Nov 12;110(46):E4385-92. doi: 10.1073/pnas.1318309110. Epub 2013 Oct 29. PMID 24170856
- [Background] Overgaard K, Werdelin L, Sorensen H, Mogensen P, Boysen G. Cytotoxic activity in plasma from patients with amyotrophic lateral sclerosis. Neurology. 1991 Jun;41(6):925-7. doi: 10.1212/wnl.41.6.925. PMID 2046943
- [Background] Pinter MJ, Waldeck RF, Wallace N, Cork LC. Motor unit behavior in canine motor neuron disease. J Neurosci. 1995 May;15(5 Pt 1):3447-57. doi: 10.1523/JNEUROSCI.15-05-03447.1995. PMID 7751923
- [Background] Roisen FJ, Bartfeld H, Donnenfeld H, Baxter J. Neuron specific in vitro cytotoxicity of sera from patients with amyotrophic lateral sclerosis. Muscle Nerve. 1982 Jan;5(1):48-53. doi: 10.1002/mus.880050109. PMID 7057805
- [Background] Conradi, S. Cytotoxic factor in plasma from ALS patients provokes haemolysis of normal erythrocytes. Acta Neurologica Scandinavica, 65: 246-247, 1982
- [Background] Ronnevi LO, Conradi S. Increased fragility of erythrocytes from amyotrophic lateral sclerosis (ALS) patients provoked by mechanical stress. Acta Neurol Scand. 1984 Jan;69(1):20-6. doi: 10.1111/j.1600-0404.1984.tb07775.x. PMID 6702416
- [Background] Ronnevi LO, Conradi S, Karlsson E, Sindhupak R. Nature and properties of cytotoxic plasma activity in amyotrophic lateral sclerosis. Muscle Nerve. 1987 Oct;10(8):734-43. doi: 10.1002/mus.880100810. PMID 3683447
- [Background] Sta M, Sylva-Steenland RM, Casula M, de Jong JM, Troost D, Aronica E, Baas F. Innate and adaptive immunity in amyotrophic lateral sclerosis: evidence of complement activation. Neurobiol Dis. 2011 Jun;42(3):211-20. doi: 10.1016/j.nbd.2011.01.002. Epub 2011 Jan 8. PMID 21220013
- [Background] Tsuboi Y, Yamada T. Increased concentration of C4d complement protein in CSF in amyotrophic lateral sclerosis. J Neurol Neurosurg Psychiatry. 1994 Jul;57(7):859-61. doi: 10.1136/jnnp.57.7.859. PMID 8021681
- [Background] Wolfgram F, Myers L. Amyotrophic lateral sclerosis: effect of serum on anterior horn cells in tissue culture. Science. 1973 Feb 9;179(4073):579-80. doi: 10.1126/science.179.4073.579. PMID 4119685
- [Background] Woodruff TM, Costantini KJ, Crane JW, Atkin JD, Monk PN, Taylor SM, Noakes PG. The complement factor C5a contributes to pathology in a rat model of amyotrophic lateral sclerosis. J Immunol. 2008 Dec 15;181(12):8727-34. doi: 10.4049/jimmunol.181.12.8727. PMID 19050293
- [Background] Pun S, Santos AF, Saxena S, Xu L, Caroni P. Selective vulnerability and pruning of phasic motoneuron axons in motoneuron disease alleviated by CNTF. Nat Neurosci. 2006 Mar;9(3):408-19. doi: 10.1038/nn1653. Epub 2006 Feb 12. PMID 16474388
- [Background] Miller RG, Mitchell JD, Moore DH. Riluzole for amyotrophic lateral sclerosis (ALS)/motor neuron disease (MND). Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD001447. doi: 10.1002/14651858.CD001447.pub3. PMID 22419278
- [Background] Pittock SJ, Lennon VA, McKeon A, Mandrekar J, Weinshenker BG, Lucchinetti CF, O'Toole O, Wingerchuk DM. Eculizumab in AQP4-IgG-positive relapsing neuromyelitis optica spectrum disorders: an open-label pilot study. Lancet Neurol. 2013 Jun;12(6):554-62. doi: 10.1016/S1474-4422(13)70076-0. Epub 2013 Apr 26. PMID 23623397
- [Background] Armitage P BG. Statistical Methods for Medical Researchers. Blackwell1994.
- [Derived] Kjaeldgaard AL, Pilely K, Olsen KS, Lauritsen AO, Pedersen SW, Moller K, Garred P. Amyotrophic lateral sclerosis and the innate immune system: protocol for establishing a biobank and statistical analysis plan. BMJ Open. 2020 Aug 5;10(8):e037753. doi: 10.1136/bmjopen-2020-037753. PMID 32759248